CLINICAL TRIAL: NCT04646382
Title: Evaluation of the Effect of Consuming a Mixture of Concentrated Allium Extracts on LDL Cholesterol Levels in Healthy Volunteers With Elevated LDL Cholesterol Levels
Brief Title: Effect of a Mixture of Allium Extracts on LDL Cholesterol Levels Volunteers With Elevated LDL Cholesterol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DOMCA S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C003
Record Dates: First submitted 2020-10-22; First posted 2020-11-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2021-11

CONDITIONS: Cardiovascular Health
Keywords: Garlic; Onion; LDL cholesterol; Cardiovascular health
MeSH Terms: interventions — Excipients

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, double-blind, parallel group nutritional intervention study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each volunteer is assigned a "participant number" that will be associated with a pot that will have all the product for the study.
  The "pot number" is the same as the "participant number".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Microcrystalline cellulose (9892- Capsules®) up to 400 mg.
  Interventions: Dietary Supplement: Garlic and onion concentrate; Dietary Supplement: Control
- Intervention (Experimental): Garlic concentrated extract. Onion concentrated extract. Microcrystalline cellulose (9892- Capsules®) up to 400 mg.
  Interventions: Dietary Supplement: Garlic and onion concentrate; Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Garlic and onion concentrate — Garlic extract concentrate (equivalent to 2 garlic cloves) and onion extract concentrate (equivalent to 1 onion).
  Other Names: AlioCare
Dietary Supplement: Control — Microcrystalline cellulose
  Other Names: Excipient

SUMMARY:
To evaluate the efficacy of daily consumption of a combination of concentrated extracts of garlic (Allium sativum L.) and onion (Allium cepa L.) on LDL cholesterol levels in healthy volunteers. Parameters related to metabolic syndrome, cardiovascular health and the immune system will also be analyzed.

DETAILED DESCRIPTION:
It is a controlled, randomized, double-blind, parallel-group nutritional intervention study.

64 healthy volunteers lwith elevated LDL cholesterol levels but who do not require pharmacological treatment will be randomly distributed into 2 equal groups: control group and intervention group.

For 8 weeks the volunteers will take the product immediately after lunch. During that time they will maintain their lifestyle and nutritional habits.

Blood samples will be taken at 0, 2, 4 and 8 weeks. Anthropometric parameters and health-related data were also measured.

Parameters related to lipid metabolism, metabolic syndrome and the immune system will be analized.

ELIGIBILITY:
Inclusion Criteria:

* LDL-cholesterol levels between 100 and 190 mg/dL.
* Freely agree to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Be pregnant.
* Have planned to change lifestyle and / or dietary habits.
* Having diabetes.
* Having a cerebrovascular disease.
* Having a serious illness.
* Taking products or drugs to control cholesterol levels or with antioxidant activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
LDL | 8 weeks.
  Serum LDL cholesterol

SECONDARY OUTCOMES:
Cholesterol | 8 weeks
  Serum total cholesterol
HDL | 8 weeks
  Serum HDL cholesterol
Triglycerides | 8 weeks
  Serum triglycerides
Glucose | 8 weeks
  Serum glucose
(untitled outcome) | 8 weeks
  Nitric oxide in serum
CRP | 8 weeks
  C-reactive protein in serum
Oxidized LDL cholesterol | 8 weeks
  Oxidized LDL cholesterol in plasma
MDA | 8 weeks
  Malondialdehyde in plasma
TAC | 8 weeks
  Plasma total antioxidant capacity
Selenium | 8 weeks
  Serun selenium
Selenoprotein P | 8 weeks
  Selenoprotein P in plasma
VCAM-1 | 8 weeks
  Endothelial adhesion molecules VCAM-1 in plasma
ICAM-1 | 8 weeks
  Endothelial adhesion molecules ICAM-1 in plasma
IL1 beta in plasma | 8 weeks
  Interleukin-1 beta in plasma
IL 6 | 8 weeks
  Interleukin-6 in plasma
IL 10 | 8 weeks
  Interleukin-10 in plasma
BMI | 8 weeks
  Body mass index (height/weight ratio)
Abdominal perimeter | 8 weeks
  Abdominal perimeter in centimeters
Blood pressure | 8 weeks
  Systolic pressure and diastolic pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Quesada, MD, Principal Investigator — Endocrinology and Nutrition Clinic of Dr. Miguel Quesada
Locations (1):
- Domca Sau, Alhendín, Granada, Spain